CLINICAL TRIAL: NCT03806738
Title: Enhancing Shared Decision-Making in Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: American Cancer Society, Inc. (Other); Carevive Systems, Inc. (Industry)
Responsible Party: Principal Investigator, Gabrielle Rocque, Assistant Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 427 BC SDM
Record Dates: First submitted 2019-01-14; First posted 2019-01-16 (Actual); Last update posted 2023-01-05 (Actual); Status verified 2023-01

CONDITIONS: Shared Decision Making
Keywords: Metastatic Breast Cancer; Treatment Decision Making; Shared Decision Making
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: Patients randomized to the intervention arm will receive the intervention-specific Carevive questionnaire, which includes standard questions with additional decision-making questions. These surveys will be repeated every 6 months until the patient has received a TP.
  Patients randomized to standard of care will receive their standard-of-care Carevive questionnaire used to generate TPs at time of enrollment and then every 6 months until a treatment decision is made.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Shared Decision Making Questionnaire (Experimental): * Patients randomized to the intervention arm will receive the intervention-specific Carevive questionnaire, which includes standard questions with additional decision-making questions. These surveys will be repeated every 6 months until the patient has received a TP.
  * One month or at the next visit following the decision, the patient will be asked to complete a research survey using REDCap.
  Interventions: Other: Intervention-specific Carevive questionnaire
- Standard of Care Questionnaire (Other): * Patients randomized to standard of care will receive the standard-of-care Carevive questionnaire used to generate TPs at time of enrollment and then every 6 months for patients with MBC who have not made a treatment decision until a treatment decision is made.
  * One month or at the next visit following the decision, the patient will be asked to complete a post-treatment survey using REDCap.
  Interventions: Other: Standard of Care questionnaire

INTERVENTIONS:
Other: Intervention-specific Carevive questionnaire — includes standard of care questions with additional decision-making questions
  Arms: Shared Decision Making Questionnaire
Other: Standard of Care questionnaire — includes the standard of care questions that are already in place for Carevive questionnaires
  Arms: Standard of Care Questionnaire

SUMMARY:
The objective of this trial is to conduct a two-arm, randomized controlled trial (RCT) of SDM Treatment Plans (TPs) delivered at the time of decision-making compared to standard oncology care (delayed delivery of standard-of-care TPs) to determine impact on SDM. The intervention will be piloted in a RCT with 140 early stage breast cancer (EBC) and 140 metastatic breast cancer (MBC) patients to assess impact. Subjects will be enrolled across two sites. Our primary outcome will be the increase in percentage of patients reporting a perception of shared decision-making.

Aim.1: The primary outcome will be to evaluate the impact of the SDM intervention on the percentage of patients perceiving shared or greater role in decision-making.

Aim 2: To evaluate the impact of the SDM intervention on provider outcomes including the percentage of providers perceiving SDM with the patient, number of treatment options offered to patients, the proportion of times that clinical trials are offered to patients, the use of NCCN guideline-based treatment, and self-report of treatment plan use.

Aim 3: Secondary fidelity and provider outcomes from audio recording will include whether providers elicit: any patient preferences during treatment planning, preferences related to physical side effects or efficacy, or preferences related to other aspects of the patient experience. We will also assess whether providers use the TP in the decision-making discussion and whether providers discuss or offer clinical trials to the patient.

DETAILED DESCRIPTION:
Two sites (UAB and MCI) will conduct the RCT of 140 patients with MBC and 140 patients with EBC comparing use of SDM TPs delivered during decision-making visits compared to TPs delivered post-decision-making. The Carevive Care Planning System (CPS) treatment planning software will be used at all clinical sites to provide treatment care plans to patients with breast cancer. This software platform, which is currently utilized after decision-making, will be modified within this project to facilitate SDM through the creation of a SDM TP utilized during decision-making. Together, the patients and physician will be able to review the patient's decision-making style, patient's desire for prognostic information treatments, and patient preferences about decision-making.

Participants will be compensated in the form of a $20 gift card at the time of consent. After the patient provides consent, the research coordinator will evaluate the electronic medical record (EMR) for completion of standard of care elements necessary for the generation of TPs. At UAB, an embedded form with the necessary information for TP generation is completed in the EMR as part of standard of care by clinical providers. If this form has not been completed, the research coordinator may either notify the provider to initiate form completion or complete this form within the EMR to ensure availability at the time of the treatment decision. If the research coordinator completes this form, it will be reviewed by a clinical provider. The completion of the form prior to consent for patients approached by telephone will be necessary to allow new patients to receive TPs if a decision is made at their initial visit. For other sites who do not use EMR forms, the clinical information will be entered directly into the Carevive platform by either the research coordinators or clinical staff.

We will survey patients as described above on an iPad using the Carevive platform at baseline and every 6 months until a treatment decision is made (intervention or standard-of-care). Post-treatment surveys will be administered using a REDCap survey. To minimize participant burden, we will allow patients to complete surveys in-person during routine clinic visits, by telephone, or at home using an e-mailed link to the survey based on patient preference. To accommodate patients who would like to complete surveys in-person, we will allow for a 1-month window around the initial 6-month survey (for those without a treatment decision within 6 months) and a 2-week window around post-treatment survey. We will record if surveys are completed by email, telephone, or in-person.After each decision-making encounter, the physician will be asked to complete a patient-specific survey in REDCap. For standard of care patients, this will include the Control Preferences Scale. For intervention patients, the survey will include both the Control Preferences Scale and three study-specific questions about use of TP during decision-making.

ELIGIBILITY:
Inclusion Criteria:

* Women age ≥ 18
* Presence of breast cancer
* Receiving any line and type of therapy (including both standard of care and clinical trials)

Exclusion Criteria:

* Patients who are not able to read and/or speak English
* Patients who are not being offered any medical therapy (hormone therapy, chemotherapy, targeted therapy) for their breast cancer
* Patients with a life-expectancy of less than 3 months
* Patients unable to provide informed consent
* Men
* Patients who do not plan to receive treatment at UAB or MCI

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 140 (Actual)
Dates: Start 2018-12-11 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Impact of Shared Decision Making | 3 years
  Impact of the SDM intervention on the percentage of patients perceiving shared or greater role in decision-making

CONTACTS AND LOCATIONS:
Overall Officials: Gabrielle B Rocque, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rocque GB, Eltoum N, Caston NE, Williams CP, Oliver MM, Moradi L, Ingram S, Azuero A, Pisu M, Bhatia S. A randomized controlled trial of shared decision-making treatment planning process to enhance shared decision-making in patients with MBC. Breast Cancer Res Treat. 2024 Aug;206(3):483-493. doi: 10.1007/s10549-024-07304-y. Epub 2024 Jun 10. PMID 38856885